CLINICAL TRIAL: NCT05166772
Title: Efficacy and Safety of Donafenib Combine With Sintilimab and HAIC (Hepatic Artery Infusion Chemotherapy，HAIC） in the First-line Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: Donafenib Combine With Sintilimab and HAIC (Hepatic Artery Infusion Chemotherapy，HAIC）in the First-line Treatment of Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20210872
Record Dates: First submitted 2021-11-29; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; HAIC; Sintilimab; Donafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib combined with Sintilimab and HAIC (Experimental): Donafenib：200mg bid； Sintilimab：200mg Q3D； HAIC：Q3W；
  Interventions: Drug: Donafenib; Drug: Sintilimab; Other: HAIC

INTERVENTIONS:
Drug: Donafenib — 200 mg BID，oral administration will start before the first HAIC treatment.
Drug: Sintilimab — 200 mg，Q3W，Intravenous infusion will performe before HAIC treatment.
Other: HAIC — Q3W. The total number of HAIC treatments was determined by the investigator based on patient needs. Dose: Oxaliplatin 85 mg / m2 for 2h, Calcium folinate 400 mg / m2 for 2h, 5-FU 400 mg / m2 for 10min, followed by 5-FU 1200 mg / m2 for 23 hours);

SUMMARY:
The investigators design a phase IIB clinical study to explore the efficacy and safety of Donafenib combined with Sintilimab and HAIC in the first-line treatment of unresectable hepatocellular carcinoma

DETAILED DESCRIPTION:
This trial is a single-arm, non-randomized and single-center clinical study of Donafenib combined with Sintilimab and HAIC in the first-line treatment of unresectable hepatocellular carcinoma. It will estimate that 30 patients who met the study criteria will be enrolled in Tianjin Medical University Cancer Institute and Hospital and treat with Donafenib combined with Sintilimab and HAIC. The investigators will follow up and collect subjects' data monthly to evaluate the efficacy and safety of treatment, including overall survival and time to progression.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join the study and sign the informed consent;
2. Age 18 ~ 80 years old (including 80 years old), male and female;
3. Patients with hepatohcellular carcinoma diagnosed clinically or confirmed by histology / cytology according to the code for diagnosis and treatment of primary liver cancer (2019 Edition);
4. Patients with unresectable or metastatic hepatocellular carcinoma;
5. No systematic treatment. If receiving adjuvant chemotherapy after local treatment more than 12 months, and patients with disease progression or metastasis can also be included in the group;
6. The end time of the last intervention, radiotherapy and ablation should be > 4 weeks;
7. Patients who underwent hepatectomy in the past should be R0 resection, and the tumor recurrence should be more than 24 months after operation;
8. At least one assessable lesion (RECIST 1.1 criteria);
9. Expected survival time ≥ 3 months;
10. ECOG 0 ~ 1;
11. Child Pugh ≤ 7;
12. Be able to cooperate to observe adverse events;
13. Major organs are functioning normally.

    1. Hemoglobin ≥ 90 g / L;
    2. ANC ≥ 1.5 × 109/L；
    3. Platelet count ≥ 75 × 109/L；
    4. Albumin ≥ 28 g / L;
    5. Total bilirubin ≤ 2 × ULN;
    6. AST, ALT ≤ 5 × ULN；
    7. ALP ≤ 5 × ULN；
    8. Creatinine ≤ 1.5 × ULN；
    9. INR or PT ≤ 1.5 × ULN； J) APTT ≤ 1.5 × ULN。

Exclusion Criteria:

1. Fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and other components confirmed by histology / cytology in the past;
2. Have a history of malignancy other than hepatocellular carcinoma unless the following criteria are met:

   A) The patient has received possible curative treatment and there is no evidence of the disease within 5 years; B) Successful resection of basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder carcinoma, carcinoma in situ of cervix and other cancers in situ
3. Diffuse tumor lesions;
4. Tumor vascular invasion occurs in one or more of the following situations:

   1. Involving superior mesenteric vein;
   2. Involving inferior vena cava;
5. History of hepatic encephalopathy, hepatorenal syndrome, or history of liver transplantation;
6. Pleural effusion, ascites and pericardial effusion with clinical symptoms requiring drainage;
7. Central system metastasis;
8. Previous history of severe mental illness;
9. Have a disease that affects absorption, distribution, metabolism, or clearance of the drug under study (such as severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorder, etc.);
10. Previous allogeneic stem cell or parenchymal organ transplantation;
11. Previously received targeted therapy of anti VEGF and / or signal pathways such as VEGFR, RAF and MEK, such as sorafenib, renvatinib and regofinib, or immunomodulator therapy such as anti-PD-1, anti-PD-L1 and anti-CTLA-4;
12. Patients who have received other anti-tumor systemic treatment in the past, including traditional Chinese medicine with anti-tumor indications less than 2 weeks before the administration of this study, or the adverse events caused by previous treatment have not recovered to ≤ CTCAE level 1; The toxicity of previous anti-tumor treatment did not include grade 1 / 2 neurotoxicity and hair loss caused by oxaliplatin;
13. Taking drugs that may prolong QTc and / or induce tip twist transition ventricular tachycardia (TDP) or drugs that affect metabolism at the same time;
14. Previous or current congenital or acquired immunodeficiency disease;
15. Active or previously documented autoimmune disease or inflammatory disease.
16. Previous allogeneic stem cell or parenchymal organ transplantation;
17. Systemic immunosuppressive drugs were used within 2 weeks before enrollment, or systemic immunosuppressive drugs expect to be needed during the study, except for the following:

    d) Intranasal, inhalation, topical or local injection (such as intra-articular injection) of corticosteroids; e) Systemic corticosteroids with dose not exceeding 10 mg / day, prednisone or other effects; f) Prophylactic use of corticosteroids for hypersensitivity;
18. Allergy to Donafenib or similar drugs, or history of hypersensitivity to chimeric or humanized antibodies or fusion proteins, or allergy to the excipients of the study drugs;
19. Have active bleeding or abnormal coagulation function, have bleeding tendency or are receiving thrombolytic, anticoagulant or antiplatelet therapy;
20. Thrombosis or thromboembolism events occurred in the past 6 months, such as stroke and / or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc;
21. Bleeding events of esophageal or gastric varices caused by portal hypertension in the past 6 months, or any life-threatening bleeding events in 3 months;
22. Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe / unstable angina or coronary artery bypass grafting in the past 6 months, congestive heart failure (NYHA grade > 2), arrhythmias poorly controlled or requiring pacemaker treatment, and hypertension not controlled by drugs (systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg);
23. Other significant clinical and laboratory abnormalities considered by the investigator to affect safety;
24. Severe infections in the active stage or under clinical control; Active infections include:

    1. HIV1/2 is positive.
    2. HBsAg positive or HBV DNA > 2000iu/ml and abnormal liver function;
    3. HCV antibody positive or HCV RNA ≥ 103 copies/ml and abnormal liver function;
    4. Active tuberculosis;
    5. Other uncontrollable active infections (CTCAE V5.0 > grade 2);
25. Not recovered from the operation, such as unhealed incision or serious postoperative complications;
26. Pregnant or lactating women, and women or men with fertility are unwilling or unable to take effective contraceptive measures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ORR（Objective Response Rate） | 1 year
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).

SECONDARY OUTCOMES:
OS（Overall survival） | 3 years
  Overall survival is defined as time from the start of treatment until death due to any reason.
TTP（Time to progress） | 3 years
  Time to Progression (TTP) defined as the time from the date of randomization to the date of first documented radiological confirmation of disease progression.
PFS（Progress free survival） | 3 years
  PFS during the retreatment phase was assessed by the site Investigator using RECIST 1.1 and defined as the time from the date of enrollment until the date of objective disease progression or death (by any cause in the absence of progression).
DCR（Disease control rate） | 3 years
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
DOR（Duration of response） | 3 years
  DoR was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression. The time of the initial response was defined as the latest of the dates contributing toward the first visit response of CR or PR. If a patient did not progress following a response, then their DoR was censored at the PFS censoring time.
AE（Adverse events） | 3 years
  Safety as measured by number and grade of adverse events

REFERENCES:
- [Derived] Gao W, Pan ZL, Zhao XH, Yang L, Cao JB, Li DY, Zheng HJ, Liu C, Li GT, Bao X, Liu XM, Zhang WH, Zhu XL, Xiao BH, Song TQ, Li Q, Lu W, Xing WG, Zhang W. Donafenib and sintilimab combined with hepatic arterial infusion chemotherapy for unresectable hepatocellular carcinoma: a prospective, single-arm phase II trial (DoHAICs study). EClinicalMedicine. 2025 May 5;83:103217. doi: 10.1016/j.eclinm.2025.103217. eCollection 2025 May. PMID 40475000